CLINICAL TRIAL: NCT02883166
Title: Improving Bio-availability of the Expensive Oral Oncolytic Drug Abiraterone by Food Intake
Acronym: SNACK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UMCN-AKF-16.04
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abiraterone; Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1 (Other): 1000mg abiraterone fasted followed by 500 mg with breakfast
  Interventions: Drug: abiraterone
- group 2 (Other): 500 mg abiraterone with breakfast followed by 1000mg fasted
  Interventions: Drug: abiraterone

INTERVENTIONS:
Drug: abiraterone — integested with a continental breakfast
  Other Names: Zytiga

SUMMARY:
Abiraterone is a selective inhibitor of androgen biosynthesis that potently and irreversibly blocks CYP17, a crucial enzyme in testosterone and estrogen synthesis. A pro-drug of abiraterone, abiraterone acetate (Zytiga®), was developed to overcome its poor bio-availability and is fully converted to the active moiety abiraterone. Abiraterone acetate tablets are administered at a fixed oral dose of 1000mg QD in a fasted state in combination with 10mg prednisolon daily.

Abiraterone acetate has a low solubility in aqueous media and a low permeability. The bioavailability of abiraterone acetate is significantly influenced when ingested with food. Ingesting abiraterone acetate with a low fat or a high fat meal resulted respectively in a 5- or 10-fold increase in AUC0-∞. The high and low fat FDA meals used in these food effect studies differ largely from breakfasts taken in everyday life (ca. 800-1000 cal). A continental breakfast contains 160 to 320 calories of which 25-50% is fat, is more compatible with a normal lifestyle and therefore easily sustainable in daily practice. However, the effect of a continental breakfast on the absorption of abiraterone is unknown yet. Furthermore, increasing healthcare costs are a growing concern in all developed countries. Therefore effort should be invested to keep anticancer treatment affordable. A food intervention resulting in a better absorption and enhanced exposure to abiraterone, can lead to a reduced dose, which could significantly impact health care costs for a tumor which is as prevalent as metastatic prostate cancer.

Therefore the investigators want to perform a bioequivalent study to investigate what dose of abiraterone with a continental breakfast equals the dose of 1000mg taken in fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow-up.

Note: informed consent may be obtained prior to start of the specified screening window.

Note: procedures conducted as part of the subject's routine clinical management (e.g. blood count) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol.

* ≥ 18 year old men who use or will start with abiraterone.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Feasible to collect blood samples from.

Exclusion Criteria:

* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:
* Malabsorption syndrome.
* Major resection of the stomach or small bowel.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Unable or unwilling to discontinue use of prohibited medications listed in APPENDIX 3 for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of day 1 and for the duration of the study.
* Concurrent use of other substances known or likely to interfere with the pharmacokinetics of abiraterone.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
dose finding | 1.5 year
  determine the equivalent dose of abiraterone when taken with a continental breakfast compared to 1000mg in fasted state

CONTACTS AND LOCATIONS:
Overall Officials: David Burger, PhD, Study Chair — Radboud University Medical Center
Locations (1):
- Radboud UMC, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lubberman FJE, Benoist GE, Gerritsen W, Burger DM, Mehra N, Hamberg P, van Oort I, van Erp NP. A prospective phase I multicentre randomized cross-over pharmacokinetic study to determine the effect of food on abiraterone pharmacokinetics. Cancer Chemother Pharmacol. 2019 Dec;84(6):1179-1185. doi: 10.1007/s00280-019-03952-w. Epub 2019 Sep 12. PMID 31515667
- See also: paper — https://link.springer.com/article/10.1007/s00280-019-03952-w